CLINICAL TRIAL: NCT06334107
Title: Mitochondrial DNA Signatures of Poor Aerobic Exercise Trainability in Young Adults Born Preterm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 24AIREA1191995
Record Dates: First submitted 2024-03-18; First posted 2024-03-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Aerobic capacity trainability; mitochondrial DNA; heteroplasmy; mitochondrial oxidative capacity
MeSH Terms: conditions — Premature Birth | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Training (Experimental): Participants will be asked to complete a 16-week aerobic exercise training program.
  Interventions: Behavioral: Exercise
- Mitochondrial DNA Sequencing (No Intervention): Participants will be asked to provide a blood or saliva sample for mitochondrial DNA sequencing analysis to assess for variants unique to individuals born prematurely.

INTERVENTIONS:
Behavioral: Exercise — Participants will be asked to follow a moderate-intensity aerobic exercise training program for 4-5 days per week for 40-60 minutes each session.
  Arms: Aerobic Exercise Training

SUMMARY:
Young adults born very preterm (32 weeks gestation or earlier) do not respond well to aerobic exercise training, meeting the recommendations set by the Physical Activity Guidelines for Americans, where they do not increase their fitness level (or cardiorespiratory fitness). Thus, they do not receive the health benefits of exercise. Achieving physical fitness through aerobic exercise training is the most cost-effective method for preventing and treating many diseases. Young adults born very preterm also have a higher risk of these conditions. Thus, their inability to respond to increase their fitness is a major problem.

One likely explanation for poor exercise trainability and increased heart disease risk in young adults born very preterm is the effect of the early birth on the major energy producers in all our cells: Mitochondria. During late-stage gestation, mitochondria change from relying on sugar as a major fuel source to fat. Unfortunately, individuals born very preterm miss this transition in fuel source reliance, which causes significant stress and damage to mitochondria. Mitochondria are critical for post-natal organ development; thus, it is thought that preterm birth-induced mitochondrial dysfunction is the underlying cause of poor trainability and high disease risk in young adults born very preterm. Indeed, mitochondrial dysfunction is evident in these individuals.

To date, there is not a way to help young adults born preterm improve their fitness level. One likely target is in the mitochondria: it's DNA. Mitochondrial DNA helps determine how mitochondria function and can be damaged under stress. Our goal in this proposed work is to determine the role of mitochondrial DNA in mitochondrial dysfunction and its link to their poor trainability.

Questions:

1. Are there mitochondrial DNA markers linked to mitochondrial dysfunction and poor exercise trainability in young adults very born preterm?
2. Do mitochondrial DNA in young adults born very preterm respond differently to aerobic exercise training than those born at term?

The investigators expect this work will show mitochondrial DNA changes linked to mitochondrial dysfunction and poor trainability, which can be used for future targets to improve health. This work supports AHA mission by helping to identify a marker in individuals born very preterm linked to their higher heart disease risk and death early in life.

DETAILED DESCRIPTION:
Young adults born very preterm (VPTB; ≤ 32 weeks gestational age) have an impaired response to aerobic exercise training (AET), often characterized by no change in aerobic capacity (VO2max) following AET. This diminishes the potential of AET to offset their elevated cardiovascular disease risk early in life VPTB's poor trainability is linked to their known mitochondrial dysfunction, thought to occur due to blunted mitochondrial maturation with early birth. Currently, no therapeutics are available to improve VO2max trainability for this population.

Data from our lab in humans and mice demonstrate that mitochondrial DNA (mtDNA) variants and other mitochondrial genomic aspects have a role in VO2max trainability. In humans, the investigators found that individuals with the largest increase in VO2max following AET had a higher occurrence of mitochondrial heteroplasmy (a shift in sequence across mtDNA). In contrast, heteroplasmy decreased in those with little-to-no change in VO2max. The reduction in heteroplasmy correlated with higher mtDNA lesions, suggesting exercise was inflicting excessive oxidative stress on mitochondria in these individuals. The investigators also identified 13 mtDNA variants in those with poor trainability, possibly linked to their lowered heteroplasmy response after exercise training. These data indicate that genetic diversity characterized by the response of mtDNA heteroplasmy with AET is an important factor determining the adaptability of VO2max with AET. To date, VPTB mitochondrial genomes have not been characterized. An onset of variants in their mitogenomes due to early birth would be easily identifiable compared to their birth mother, given that mtDNA is maternally inherited. Importantly, these mitogenome variants may inform the effect of AET on heteroplasmy and their low trainability. Thus, there is a critical need to characterize VPTB mitochondrial genome characteristics and how AET influences these dynamics.

Our long-term goal is to improve mitochondrial function and VO2max trainability in VPTB young adults facing disproportionately higher disease risk where exercise is known to be beneficial as a treatment and preventative measure. Accordingly, the overall objectives of this application are to i) characterize VPTB-induced mtDNA changes in sequence, heteroplasmy, and damage, and ii) determine the effect of AET on these mtDNA traits and mitochondrial function in cells known to correlate with heart mitochondrial oxidative capacity: namely peripheral blood mononuclear cells (PBMCs). Our central hypothesis is that VTPB young adults will have unique mtDNA variants/mutations and that AET will significantly decrease PBMC mtDNA heteroplasmy and copies alongside lowered mitochondrial oxidative capacity compared to normal-term birth (NTB) adults. The rationale for this project is that characterizing unique VPTB mtDNA aspects and the heteroplasmy response to AET might reveal an underlying mechanism for their poor trainability that can be targeted for future work. To meet these objectives, the investigators will assess these two specific aims: Aim 1: Assess for informative mtDNA variants in VPTB young adults. The investigators hypothesize there will be de novo mtDNA variants in VPTB offspring compared to their birth mothers.

Aim 2: Determine the effect of AET on mitochondrial oxidative capacity and mtDNA heteroplasmy, copy number, and lesions in isolated PBMCs in VPTB and NTB young adults. The investigators hypothesize VPTB adults will exhibit decreased mtDNA heteroplasmy and increased lesions following AET compared to age-matched NTB adults.

After completing the proposed research, our expected outcome is identifying a unique signature of mtDNA variants and heteroplasmy responses to AET in VPTB adults that will explain their low trainability. These results are expected to have a positive impact for researchers because it will provide a foundation for future research to target mtDNA as a strategy to help VPTB adults reduce their risk for cardiovascular disease and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Preterm born (PTB)young adult group: Participants must be inactive (reported exercise < 150 mins/week; See IPAQ Attachment), males and females aged 18-35 years born preterm with a gestational age <37 weeks.
* Normal term-born (NTB) young adult control group: Participants must be inactive (reported exercise < 150 mins/week) and will be age- and sex-matched and born at term (37 gestational age).
* The biological mother of PTB participants: The PTB biological birth mother must be the one who gave birth to the participant and the one from whom the child inherited half of its genetic background (i.e., DNA).
* PTB and NTB young adults must pass the PAR-Q+ Questionnaire assessment, indicating readiness to begin a moderate-intensity exercise training program. We will follow the American College of Sports Medicine's aerobic exercise training program participation guidelines. Subjects who are cleared via the PAR-Q+ assessment will be permitted to participate in the training program.

Exclusion Criteria:

• PTB and NTB young adults only: Having a diagnosed bronchopulmonary hyperplasia, cardiovascular (cardiac or peripheral arterial disease), metabolic (Diabetes Mellitus Type 1 or 2), or renal or liver disease, and signs or symptoms of these conditions, including pain: discomfort in the chest, neck, jaw, arms, or other areas that may result from ischemia; shortness of breath at rest or with mild exertion; dizziness or syncope; orthopnea or paroxysmal nocturnal dyspnea; ankle edema; palpitations or tachycardia; intermittent claudication; known heart murmur; unusual fatigue or shortness of breath with usual activity.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial DNA heteroplasmy | Immediately after aerobic exercise training intervention; change in pre- to post-frequency
  The full-length mitochondrial DNA sequence will be analyzed and assessed for heteroplasmic sites in the mitochondrial genome. Briefly, mitochondrial DNA exists in many copies, and heteroplasmy is noted when the amino acid sequence changes from the major read 2% or more across the DNA copies. The change in the mean heteroplasmy frequency and the mean number of sites with heteroplasmy with aerobic exercise training by comparing these changes in young adults born preterm to those born at term.
Mitochondrial DNA sequence variants | Immediately after visit 1
  The full-length mitochondrial DNA sequence will be determined in participants who report being born prematurely, which will be compared to their biological birth mother. In this comparison, we will assess for variants. We deem a site as an 'informative' mitochondrial DNA variant in young adults born prematurely as a change in amino acid sequence from the biological birth mother.
Change in maximal aerobic capacity | Immediately after aerobic exercise training intervention; change in pre- to post-frequency
  The change in maximal aerobic capacity will be assessed via the modified Balke-graded exercise test before and after the aerobic exercise training program.
Change in mitochondrial oxidative capacity in peripheral blood mononuclear cells | Immediately after aerobic exercise training intervention; change in pre- to post-frequency
  Mitochondrial maximal respiration (i.e., oxidative capacity) will be measured in isolated peripheral blood mononuclear cells.

SECONDARY OUTCOMES:
Daily sleep habits | Daily for 16 weeks.
  Daily sleep data will be collected from the Fitbit Charge via the Fitabase software program during the experimental period. Subjects will be instructed to create a habit of wearing their Fitbit Charge each night of the training period. At the completion of the study, the research team will collect daily sleep data that includes the estimated time spent (i.e., minutes or seconds) in each stage (awake, rapid eye movement, light, and deep).

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University | Kinesiology and Sport Management Building, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT06334107/Prot_SAP_000.pdf